CLINICAL TRIAL: NCT02273804
Title: Topiramate and Severe Obesity in Children and Adolescents
Brief Title: Topiramate and Severe Obesity
Acronym: TOBI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P091122; 2011-006193-36 (EudraCT Number)
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Obese Children and Adolescents
Keywords: Topiramate; Obesity; Children; Adolescents
MeSH Terms: conditions — Obesity | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- topiramate (Experimental): pill
  Interventions: Drug: Topiramate
- placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate for 9 months treatment, and then 27 months of follow-up Dose regimen will be determined according to theoretical weight (taken orally), escalated every 15 days. Patients who do not tolerate dose escalation will be reduced to the highest tolerated dose.
  Arms: topiramate
Drug: Placebo — Placebo will be taken orally following to the same dose regimen according to theoretical weight
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of Topiramate on the decrease of Body Mass Index compared to placebo at 9 months.

DETAILED DESCRIPTION:
Childhood obesity remains through adulthood in main cases, and is associated with an early increase of cardiovascular risk and an excess mortality in young adults due to stroke and cancer.

Bariatric surgery is very rare in France for children and can cause severe complications. Long term effects are still unknown.

Topiramate is already use in thousands of children in neurology, its effects are already well known, and no lethal complication is reported.

The hypothesis is that Topiramate associated with standard treatment of obesity is more effective than standard treatment alone.

This will be a 4.5-years, randomized, double-blind, placebo-controlled, clinical trial of topiramate (9 months) vs placebo (9months) for Body Mass Index reduction in 160 adolescents (ages 9-17 years old) with severe obesity.

The main objective is to evaluate the efficacy of Topiramate on the decrease of Body Mass Index compared to placebo at 9 months.

The secondary objectives are to evaluate:

* the decrease of Body Mass Index Z-score
* the tolerance of Topiramate
* the effectiveness of Topiramate on weight decrease and decrease of Body Mass Index and Body Mass Index Z-score at 1, 3 ,4 and 6 months
* the effectiveness of Topiramate on eating behaviour, physical activity, calculated with validated questionnaires and scales at 6 and 9 months
* the pharmacokinetic of Topiramate in obese children and adolescents

ELIGIBILITY:
Inclusion Criteria:

* 9-17 years old
* Body Mass Index Z-score ≥ 4 SD of French reference
* Weight at enrolment ≥ 50 kg
* Therapeutic failure > 6 months
* For girls of childbearing age, willing to have an acceptable method of contraception (no estrogens plus progestin)
* Negative pregnancy test for girls of childbearing age
* Agreeing to participate upon written informed consent
* Appropriate understanding of the study

Exclusion Criteria:

* Syndromic or secondary obesity
* Major neurological or psychiatric disorder
* Current or history of suicidal thought/attempts
* Current or history of breakdown
* Previous bariatric surgery
* Severe hypercapnia
* Renal dysfunction
* Deformity in the urinary tract or solitary kidney
* History of renal lithiasis or glaucoma
* Poorly controlled diabetic children or adolescents (HbA1c >10%) and diabetic patients treated with Metformine and/or glibenclamide
* Hepatic dysfunction
* Bicarbonate ≤16 mmol/L
* Known hypersensitivity to the active substance or to one of the excipients
* Intolerance to saccharose
* Enrolment in another therapeutic study
* High probability to fail to comply with treatment
* Females: Pregnant, planning to become pregnant
* No signature on consent form
* Uncovered by the French National health Insurance system (Sécurité sociale)

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Mass Index (BMI) | 9 months
  Success is defined by a percent change > 2.5%

SECONDARY OUTCOMES:
Adverse event outcome | Up to 4,5 years of follow-up
Percent Change from Baseline in Body Mass Index Z-score | 9 months
Percent Change from Baseline in Body Mass Index and Body Mass Index Z-score | 1 months
Percent Change from Baseline in Body Mass Index and Body Mass Index Z-score | 3 months
Percent Change from Baseline in Body Mass Index and Body Mass Index Z-score | 4 months
Percent Change from Baseline in Body Mass Index and Body Mass Index Z-score | 6 months
Eating Behaviour | 6 months
  Self-administered questionnaires and scales :
  Binge Eating Scale ; State trait anxiety Inventory for Children; Child depression inventory, Child Behavior Checklist
Eating Behaviour | 9 months
  Self-administered questionnaires and scales :
  Binge Eating Scale ; State trait anxiety Inventory for Children; Child depression inventory; Child Behavior Checklist
Physical activity | 6 months
  Questionnaire from French Ministry of Health
Physical activity | 9 months
  Questionnaire from French Ministry of Health
Food intake | 6 months
  High-fat, sugary, salted food intake and beverage other than drinking water
Food intake | 9 months
  High-fat, sugary, salted food intake and beverage other than drinking water
Comorbidity outcome | 6 months
  Comorbidities and metabolic and cardiorespiratory complications
Comorbidity outcome | 9 months
  Comorbidities and metabolic and cardiorespiratory complications

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Frelut, MD, Study Chair — Assistance Publique - Hôpitaux de Paris; Gianpaolo De Filippo, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bicêtre, Le Kremlin-Bicêtre, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGovern L, Johnson JN, Paulo R, Hettinger A, Singhal V, Kamath C, Erwin PJ, Montori VM. Clinical review: treatment of pediatric obesity: a systematic review and meta-analysis of randomized trials. J Clin Endocrinol Metab. 2008 Dec;93(12):4600-5. doi: 10.1210/jc.2006-2409. Epub 2008 Sep 9. PMID 18782881
- [Background] Bray GA. Risks of obesity. Endocrinol Metab Clin North Am. 2003 Dec;32(4):787-804, viii. doi: 10.1016/s0889-8529(03)00067-7. PMID 14711062
- [Background] Astrup A, Caterson I, Zelissen P, Guy-Grand B, Carruba M, Levy B, Sun X, Fitchet M. Topiramate: long-term maintenance of weight loss induced by a low-calorie diet in obese subjects. Obes Res. 2004 Oct;12(10):1658-69. doi: 10.1038/oby.2004.206. PMID 15536230
- [Background] Toplak H, Hamann A, Moore R, Masson E, Gorska M, Vercruysse F, Sun X, Fitchet M. Efficacy and safety of topiramate in combination with metformin in the treatment of obese subjects with type 2 diabetes: a randomized, double-blind, placebo-controlled study. Int J Obes (Lond). 2007 Jan;31(1):138-46. doi: 10.1038/sj.ijo.0803382. Epub 2006 May 16. PMID 16703004
- [Background] Rosenstock J, Hollander P, Gadde KM, Sun X, Strauss R, Leung A; OBD-202 Study Group. A randomized, double-blind, placebo-controlled, multicenter study to assess the efficacy and safety of topiramate controlled release in the treatment of obese type 2 diabetic patients. Diabetes Care. 2007 Jun;30(6):1480-6. doi: 10.2337/dc06-2001. Epub 2007 Mar 15. PMID 17363756